CLINICAL TRIAL: NCT02264769
Title: Carbetocin at Elective Cesarean Deliveries: A Non-inferiority Study Between 20 and 100 Micrograms - Part 4
Brief Title: Carbetocin at Elective Cesarean Delivery Part 4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-03
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Postpartum Hemorrhage
Keywords: pregnancy; postpartum hemorrhage; Cesarean delivery; carbetocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbetocin 20mcg (Active Comparator): Patient is given carbetocin 20 mcg intravenously over 1 minute, immediately upon delivery of the anterior shoulder of the baby.
  Interventions: Drug: Carbetocin
- Carbetocin 100mcg (Active Comparator): Patient is given carbetocin 100 mcg intravenously over 1 minute, immediately upon delivery of the anterior shoulder of the baby.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin
  Other Names: Duratocin

SUMMARY:
PostPartum hemorrhage (PPH) is a major cause of maternal death worldwide. Oxytocin is the most commonly used uterotonic drug to prevent and treat PPH in North America. However oxytocin has a very short duration of action, requiring a continuous infusion to achieve sustained uterotonic activity. Moreover large doses are associated with adverse effects like hypotension, nausea, vomiting, dysrhythmias and ST changes. The Society of Obstetricians and Gynecologists of Canada (SOGC) has recommended a single dose of 100 mcg of carbetocin at elective cesarean delivery to promote uterine contraction. In three studies recently performed at Mount Sinai Hospital, the investigators have found no difference in uterine contractility between the doses of 20- 120 mcg carbetocin and that the ED90 is 14.8 mcg. Thus a larger trial comparing the minimum effective dose determined in the previous three trials with the standard 100 mcg dose is necessary to confirm these findings.

DETAILED DESCRIPTION:
The current oxytocin regimen requires the administration of a continuous infusion to achieve sustained uterotonic activity, which can be associated with a number of side effects and unpredictable efficacy. Carbetocin in a single 100 mcg dose has apparently greater efficacy, with a similar side effect profile to that of oxytocin. In addition, some studies have also shown that there is less blood loss and less requirement for additional uterotonic drugs when carbetocin is administered. Studies conducted by the investigators group at Mount Sinai have shown similar efficacy between the doses ranging from 20 to 100 mcg of carbetocin. In the investigators study, the investigators are going to compare those two doses of carbetocin to determine that 20 mcg is not inferior to 100 mcg to produce adequate uterine tone in elective cesarean delivery. This study will be a randomized, double - blind, non inferiority study.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean delivery under spinal anesthesia.
* Written informed consent to participate in this study.
* Term pregnancy

Exclusion Criteria:

* Refusal to give written informed consent.
* Allergy or hypersensitivity to carbetocin or oxytocin.
* Conditions that predispose to uterine atony and postpartum hemorrhage, such as placenta previa, multiple gestation, preeclampsia, eclampsia, macrosomia, polyhydramnios, uterine fibroids, previous history of uterine atony and postpartum bleeding, or bleeding diathesis.
* Hepatic, renal, and vascular disease.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Uterine tone | 2 minutes
  Uterine tone on a scale of 0-10 at 2 minutes after completion of injection of carbetocin.

SECONDARY OUTCOMES:
Uterine tone | 5 minutes
  Uterine tone on a scale of 0-10 at 5 minutes after completion of injection of carbetocin.
Additional uterotonic medication administration | 24 hours
  2. The use of additional uterotonic at any time post administration of carbetocin up to 24 hours post delivery.
Blood loss | 48 hours
  Blood loss will be calculated through the difference in hematocrit values assessed prior to and at the end of 48 hours after the cesarean section.
Side Effects | 2 hours
  Any of the following will be noted up to 2 hours post delivery: systolic blood pressure < 80% of pre-delivery values, tachycardia > 30% pre-delivery levels, bradycardia < 30% pre-delivery levels, other dysrhythmias, nausea, vomiting, chest pain, shortness of breath, headache, flushing, others

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada